CLINICAL TRIAL: NCT02736734
Title: The Effect of Corticotrophin-releasing Hormone (CRH) on Esophageal Motility in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prof Dr Jan Tack (Other)
Responsible Party: Sponsor-Investigator, Prof Dr Jan Tack, Prof. Dr., MD, PhD, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: S57111
Record Dates: First submitted 2015-12-10; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Esophageal Motility Disorders
MeSH Terms: conditions — Esophageal Motility Disorders | interventions — Corticotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CRH condition (Other): All HV first underwent a baseline manometry measurement. After 30 minutes, an intravenous CRH injection was done. The same measurement was repeated but now with CRH administered.
  Interventions: Drug: CRH

INTERVENTIONS:
Drug: CRH — CRH injection: 100 µg CRH powder for injection (CRH Ferring) dissolved in 1ml NaCl 0.9%, administration intravenously over the course of 1 minute to avoid side effects.
  Other Names: CRH, Ferring

SUMMARY:
Stress is well known to affect visceral sensitivity and gastrointestinal function in general. A majority of patients with gastroesophageal reflux disease (GERD) report stress as an important factor triggering symptom exacerbation. A real-life stressor could exacerbate heartburn symptoms in GERD patients by enhancing perceptual response to esophageal acid exposure. In Irritable Bowel Syndrome (IBS) patients, visceral hypersensitivity is a major pathophysiological mechanism and stress is shown to trigger or exacerbate symptoms.

A possible mechanism of stress-induced visceral sensitivity could be the barrier dysfunction. Indeed, in a study performed by our group, in human, an acute psychological stressor induces hyperpermeability in a mast cell dependent fashion and exogenous peripheral corticotrophin-releasing hormone (CRH) recapitulated its effects on barrier function. This increase in intestinal permeability is a phenomenon which appears as a prerequisite for visceral hypersensitivity. Furthermore, few studies indicate that human intestinal motility is probably modulated by CRH. It has been shown that the brain-gut axis in IBS patients has an exaggerated response to CRH.To our knowledge, the acute effect of exogenous CRH on esophageal motility has not been studied before.

DETAILED DESCRIPTION:
1. INTRODUCTION Gastro-esophageal reflux disease (GERD), defined as the presence of symptoms or lesions that can be attributed to the reflux of gastric contents into the esophagus, is an increasingly prevalent condition in Western societies. The most typical symptoms are heartburn and regurgitation, but GERD can manifest itself through a variety of esophageal and extra-esophageal symptoms (e.g. chronic cough).

   In humans, pain is a multimodal experience composted of sensory, physiological and psychological aspects. In order to mimic the clinical situation, experimental models should be based on testing regimens in which different receptors and central nervous system mechanisms are activated.

   Advances in esophageal sensory stimulation have established that both typical and atypical symptoms may not only arise from acid reflux, but also from reflux events with less acidic pH (pH 4-7). In GERD patients with symptoms that persist in spite of acid suppressive therapy, ongoing weakly-acidic and non-acid reflux is now well established as the main underlying factor.

   The basis for symptom generation during weakly-acidic reflux events remains to be determined, but acid sensitivity in the pH range 4-7, mechanical distention (enhanced by air in the refluxate), sensitivity to other chemical factors (e.g. bile) and esophageal hypersensitivity to physiological levels of reflux have all been proposed.

   The investigators speculate that visceral hypersensitivity plays an important role in symptom perception. This is suggested by the reflux parameters that are usual within the physiological number during proton pump inhibitor (PPI) therapy. Also, our group previously demonstrated that refractory GERD patients have increased visceral hypersensitivity for thermal, chemical and mechanical esophageal stimulation compared to healthy volunteers.

   Stress is well known to affect visceral sensitivity and gastrointestinal function in general. A majority of patients with GERD report stress as an important factor triggering symptom exacerbation. A real-life stressor could exacerbate heartburn symptoms in GERD patients by enhancing perceptual response to esophageal acid exposure. In Irritable Bowel Syndrome (IBS) patients, visceral hypersensitivity is a major pathophysiological mechanism and stress is shown to trigger or exacerbate symptoms.

   A possible mechanism of stress-induced visceral sensitivity could be the barrier dysfunction. Indeed, in a study performed by our group, in human, an acute psychological stressor induces hyperpermeability in a mast cell dependent fashion and exogenous peripheral corticotrophin-releasing hormone recapitulated its effects on barrier function. This increase in intestinal permeability is a phenomenon which appears as a prerequisite for visceral hypersensitivity. Furthermore, few studies indicate that human intestinal motility is probably modulated by CRH. It has been shown that the brain-gut axis in IBS patients has an exaggerated response to CRH.To our knowledge, the acute effect of exogenous CRH on esophageal motility has not been studied before.
2. RATIONALE AND OBJECTIVES CRH is considered to be a prominent mediator of stress responses in the brain-gut axis. In particular, stress-related activation of CRH receptors has been reported to produce alterations in gastrointestinal function. In a first study, the investigators studied the effect of CRH on esophageal sensitivity in healthy volunteers (HV). Preliminary results demonstrated that CRH-administration increased esophageal sensitivity (pain perception threshold) to mechanical stimulation of the esophagus. In the present study the investigators want to study whether exogenous CRH changes the response to mechanical stimulation through an effect on esophageal contractility. Therefore, the aim of this study is to investigate the effect of CRH-administration on esophageal motility during a standard high resolution manometry (HRM) in HV.
3. GENERAL DESCRIPTION OF THE STUDY This study will be performed in 15 HV, to have sufficient data to compare volunteers mutual and to be able to make conclusions. All participants will sign a copy of the informed consent, attached as appendix, before initiation of the study. Esophageal motility will be measured by a standard HRM before and after administration of CRH.

   Inclusion criteria include an age between 18 to 60 years old and no history of gastrointestinal symptoms or complaints.

   Exclusion criteria include history of allergic reaction to CRH, atopy (eczema, asthma, food allergies, allergic rhinoconjunctivitis) or multiple allergies to several drugs, pregnancy or lactation, concomitant administration of monoamine oxidase inhibitors (MAOI), verapamil or diltiazem or medication affecting esophageal motility, significant co-morbidities (neuromuscular, psychiatric, cardiovascular, pulmonary, endocrine, autoimmune, renal and hepatic), prior history of esophageal, Ear Nose and Throat (ENT) or gastric surgery or endoscopic anti-reflux procedure, history of gastrointestinal disease and first degree relatives with Crohn's disease or celiac disease. During the last two weeks before the study, HV should be free from medication, except for oral contraceptives.

   Each subject that is willing to participate in this study will be submitted to a physical examination. Medical history will be taken and the use of medication will be inquired.
4. MATERIALS AND METHODS High Resolution Manometry Esophageal body pressure, peristalsis and pressure of the lower esophageal sphincter (LES) and the upper part of the stomach will be measured using HRM, as it is routinely performed in the university hospital of Gasthuisberg in patients with symptoms of dysphagia. HRM consists of measuring multiple pressures simultaneously and this allows detailed assessment of all relevant data for the entire esophagus.

CRH administration The effect of CRH-administration on esophageal motility will be studied. After positioning of the HRM probe the investigators will first study esophageal motility at baseline conditions. After the baseline procedure, 100µg CRH powder for injection (CRH ferring®, Ferring, Aalst, Belgium) will be dissolved in 1 mL of sodium chloride (NaCl) 0.9%, the solution will be injected intravenously over the course of 1 minute. With this dose, the side-effects are limited to transient facial flushing that lasts from 5 to 45 minutes in 75% of patients. CRH is clinically used as a diagnostic tool in locating the source of hypercortisolism in Cushing's disease. After 20 minutes, esophageal peristalsis will be studied again.

Saliva Samples Salivary samples will be obtained during the HRM procedure and will be used to determine salivary cortisol at baseline conditions, immediately before the CRH-administration, 30 minutes and 60 minutes after administration. Salivary cortisol will be determined by ELISA (DRG Diagnostics, Marburg, Germany) according to the manufacturer's instructions.

Assessment of emotional state An assessment of general mood will be performed by the Profile of Mood Schedule (POMS) and the State-Trait Anxiety Inventory (STAI state) questionnaires before and after the esophageal manometry. The POMS consists of 32 pairs of words that describe different feelings and emotions at the present moment. The STAI state is validated, and widely used questionnaire measuring transitory anxiety states. The scale consists of 20 items, which are answered on a 4-point scale. Scores are expressed as total sum scores.

PROTOCOL After an overnight fast volunteers will come to the endoscopy unit of the UZ Gasthuisberg, where the study will be performed. At the beginning of the study, the solid-state manometric catheter consisting of 36 manometry channels at 1cm intervals and 16 impedance channels (Medical Measurement Systems, Enschede, The Netherlands) will be placed transnasally under topical anesthesia and will be positioned along the esophagus. Manometry will measure pressure in the esophageal body, and the LES and the upper part of the stomach. The impedance channels are used to measure bolus movement. After the catheter is positioned in the esophagus the volunteer will remain in a bed, in semi-recumbent position for the entire study period. HRM and impedance will be recorded for approximately 2 hours.

Primarily, baseline recordings will be obtained. Test boluses of 5 mL liquid, 5 mL semisolid, and 2 cm2 solid will be administered orally. During every swallow, volunteers will be asked to complete a 5-point scale to monitor sensation of bolus hold up with 1 = normal passage, 2 = slow passage, 3 = step-by-step passage, 4 = partial blockage, and 5 = complete blockage. After the manometry at baseline conditions, CRH will be administered IV and a waiting period of 20 minutes will be taken into account since previous protocols with CRH administration showed that 20 to 30 minutes after CRH injection, salivary cortisol levels are the highest. After the waiting period we will repeat the same procedure used under baseline conditions.

ELIGIBILITY:
Inclusion Criteria:

* No history of gastrointestinal symptoms or complaints.

Exclusion Criteria:

* History of allergic reaction to CRH, atopy (eczema, asthma, food allergies, allergic rhinoconjunctivitis) or multiple allergies to several drugs
* Pregnancy or lactation
* Concomitant administration of monoamine oxidase inhibitors (MAOI), verapamil or diltiazem or medication affecting esophageal motility
* Significant co-morbidities (neuromuscular, psychiatric, cardiovascular, pulmonary, endocrine, autoimmune, renal and hepatic)
* Prior history of esophageal, Ear Nose and Throat, or gastric surgery or endoscopic anti-reflux procedure
* History of gastrointestinal disease and first degree relatives with Crohn's disease or celiac disease.
* During the last two weeks before the study the volunteers should be free from medication, except for oral contraceptives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in esophageal contractile properties after Intravenous CRH administration in Healthy Volunteers | approximately 2 hours study period, effect of CRH will be evaluated 30 minutes after the administration
  The investigators will evaluate if the administration of intravenous CRH alters esophageal contractile properties. Esophageal contractile properties are measured by high resolution manometry (HRM). HRM measurements in the esophagus will be performed before and after CRH administration. The investigators will compare 3 HRM parameters (distal contractile integral (mmHg.s.cm), intrabolus pressure (mmHg), LES relaxation (mmHg)) before and after the administration of CRH and assess the number of HV in which these 3 parameters are altered after CRH administration to be able to report changes in contractile properties of the esophagus.

CONTACTS AND LOCATIONS:
Overall Officials: Jan F Tack, MD, PhD, Principal Investigator — KU Leuven
Locations (1):
- Targid, KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No